CLINICAL TRIAL: NCT04387708
Title: Reorganization of Care in Patients Hospitalized in Child Psychiatry for Anorexia Nervosa at the Time of the Coronavirus-19 Epidemic in France: Qualitative Study Carried Out on Patients and Their Parents
Brief Title: Care in Patients Hospitalized for Anorexia Nervosa at the Time of the Coronavirus-19 Epidemic (QUALICOVID)
Acronym: QUALICOVID
Status: Completed | Type: Observational
Sponsor: Centre Psychothérapique de Nancy (Other)
Responsible Party: Sponsor
Other Study IDs: RIPH 2020-01; IDRCB 2020-A01101-38 (Other: ANSM (French competent authority))
Record Dates: First submitted 2020-05-13; First posted 2020-05-14 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2020-05

CONDITIONS: Anorexia Nervosa
Keywords: anorexia nervosa; child psychiatry; covid-19; qualitative study
MeSH Terms: conditions — Anorexia Nervosa; COVID-19

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Anorexia nervosa is a severe psychiatric condition. On the nutritional level, one of the objectives recommended by the High Authority of Health is to "achieve and maintain an appropriate weight and nutritional status". It is recommended that, in the event of hospitalisation, this should be "as long as necessary" and be based on a weight contract as a condition for discharge. Within the Pôle Universitaire de Psychiatrie de l'Enfant et de l'Adolescent of the Centre Psychothérapique de Nancy, an inpatient unit takes care of children and adolescents with a specific valence in the management of patients suffering from eating disorders.

Since the first quarter of 2020, France has been progressively affected by the pandemic of the coronavirus 2019, Covid-19. This pandemic has led to unprecedented containment measures in France and around the world.

At the time of the announcement of the implementation of containment, the investigators proposed to the parents of patients hospitalized in the Child and Adolescent Psychiatry Department of the Nancy Psychotherapy Center who were approaching their discharge weight to be able to end their hospitalization prematurely. As a follow-up to this hospitalisation, intensive outpatient care was offered to the families, in accordance with State recommendations in connection with the pandemic. In this hospitalized unit, weekly outpatient consultations were maintained and coupled with telephone interviews, teleconsultation interviews and a telephone hotline for the healthcare team.

The objective of the study is to explore, in a qualitative way, the experiences of patients hospitalized in the child psychiatry department for anorexia nervosa at the time of the coronavirus epidemic in France and those of their parents, in relation to the reorganization of care.

DETAILED DESCRIPTION:
Interviews will be recorded, made anonymous and transcribed verbatim. The resulting text will be subjected to an inductive thematic analysis. The investigators will analyse the interviews to identify themes. Then, based on the preliminary results, higher key themes will be proposed, i.e. the themes most present and salient in the material. They will look for a concordance between the different members of each family. Several profiles may be proposed based on the patient's and parents' experiences and will be presented in the form of a thematic tree.

The study will be proposed to all eligible patients in order to obtain as much material as possible.

ELIGIBILITY:
Inclusion Criteria:

* Criteria for inclusion :

  1/ For patients :
* To have been hospitalized in the child and adolescent psychiatry unit of the Pôle Universitaire de Psychiatrie de l'Enfant et de l'Adolescent du Centre Psychothérapique de Nancy on 16 March 2020
* With a diagnosis of anorexia nervosa (ICD-10 F500)
* Understand and speak French fluently
* Have been informed of the study, have received the study briefing note and have not objected to participating in the study.
* That the holders of parental authority have been informed of the study, have received the information note on the study and have not objected to their child's participation
* Be affiliated to or entitled to a social security scheme

  2/ For the parents :
* To have a child who meets the inclusion criteria mentioned above.
* Understand and speak French fluently
* Have been informed of the study, have received the study briefing note and have not objected to participating in the study.

Exclusion Criteria:

* no

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The source population represents six patients, aged 9 to 17 years in March 2020 and their parents.
  Four of the six patients went home on the day the lockdown measures were announced, one patient went home three days later so that her parents would be available, and one patient remained in hospital because of a physical condition incompatible with a return home.
  The population is therefore made up of 18 people: patients (6) and their parents (12).
  It will be possible to interview the parent(s) without interviewing the child if the child refuses to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2020-05-12 (Actual); Primary Completion 2020-05-20 (Actual); Study Completion 2020-05-20 (Actual)

PRIMARY OUTCOMES:
Content analysis concerning the reorganization of care for children or adolescent and thier parents | 1 interview for each participant during 45 minutes
  Analyzing the discourse content regarding the experiences related to changes in the care of patients with anorexia nervosa hospitalized in a child and adolescent psychiatric ward in Nancy, France, and their parents, in the context of the Covid-19 crisis.

CONTACTS AND LOCATIONS:
Overall Officials: Marilou Lamourette, MD, Principal Investigator — Centre Psychothérapique de Nancy
Locations (1):
- Centre Psychothérapique de Nancy, Laxou, France

IPD SHARING:
Plan to Share IPD: No